Increasing Teen Access to Care (AccessKCTeen2) NCT05444855 24 August 2022

## AccessKCTeen 2.0 Study Information Intervention Participant

PI: Melissa Miller; STUDY 000002100

**Who is doing this research study?** This study is being done by researchers at Children's Mercy Research Institute. Dr. Melissa Miller is leading this research study. Other health care professionals may help.

What is this research study about? We started the *AccessKCTeen 2.0* program to find out how we can work with teens and their friends to connect teens in the community to sexual and mental health. Sexual health can include information about birth control, sexually transmitted infection (STI) testing, relationships, and having sex. Mental health can include information about your worries or stressful situations. The purpose of this research study is to learn if the program helps teens get care they need.

Why am I being asked to be in this study? We are asking you to be part of this research study because you are an adolescent.

## What will I be asked to do if I decide to be in this study?

In this study, there are two groups of teens. If you choose to be in this study, everyone will be part of a friend network and some teens will be asked to be peer leaders.

Friend network: You will be asked to complete up to 4 surveys online or in-person. Each survey will take about 5-10 minutes to fill out. The surveys will ask questions like where you get healthcare, your sexual and mental health, relationships with friends, and trust in health care.

- You will take the first survey online or in-person after you agree to be in the study.
- We will call, email, or text you at 2, 4, and 6 months from today and ask you to do another survey.

Peer leader: You will be asked to complete the same surveys as above and there will be some added questions about your experience as a peer leader.

- You will be asked to invite friends to enroll in the study as part of your friend network.
- You will be asked to a training session to learn about health care and sharing health information. This will last about 3 hours and may be in-person or virtual.
- You can choose to share sexual and mental health information from our program, if you
  want. This will include information about health events we will host in the community as
  part of our program.
- You will be asked to respond to text messages or emails about how it is going with sharing health information.

There is no extra cost for being in the study.

## Turning 18:

When you reach adulthood (18 years of age), we will contact you to find out you want to give verbal consent for continued participation in this study.

If you cannot be reached or choose not to consent, the link between your identifiable information and the collected information will be destroyed. No identifiable information will be saved. The de-identified information will be kept in a using a secure data transfer system.

What are the benefits? There may not be direct benefit to being in this study. By being in this study, you may learn more about how to take care of your own health and help researchers find better ways to connect teens to health care through peer networks.

What are the risks? There is minimal risk to be in this study. You may feel uncomfortable answering questions about your sexual and mental health. You do not have to give any information you do not want to give. You may skip any questions that make you uncomfortable. There's a small risk of a breach of confidentiality (someone could find out your survey answers or what you said), and there is a risk of unsecure two-way texting. We will protect your information as much as possible, and if any information like your name, address, date of birth etc. is shared through text, a member of our team will call you.

What identifiable information will we use for this study? Information that will be collected will include your name, date of service, contact information, email address and phone number. We will work to ensure that your information is kept private. We will keep this information until the end of the study. Other people at Children's Mercy Hospitals, University of Kansas Medical Center (KUMC), and University of Missouri-Kansas City (UMKC) may look at the data we collect and may see your study information.

We will remove information that identifies you (such as your name, phone number, and email) from our data and use the rest of the data we collected for future studies without asking your permission. We may also share your non-identifying information with other researchers for future studies without asking your permission.

**How will my information be used in the future?** All survey responses will be compiled into an anonymous summary where we will share with our community partners, other Children's Mercy, KUMC, and UMKC staff. There will be no names attached to this summary. We may also share your non-identifying information with other researchers for future studies without asking your permission.

What are the alternatives to being in this study? Instead of being in this study, you may choose not to be in this study. Being in this study is completely voluntary and will not affect any care at any Children's Mercy Hospital. You may change your mind at any time. Your decision will not impact any future care you receive at Children's Mercy.

## What will I receive for being in this study?

Friend network: You can receive up to \$60 for being in this study.

- You will get \$30 for completing the first (baseline) survey.
- You will get \$10 for completing each of the follow-up surveys at 2, 4, 6 months

Peer leader: You can get the same amount (\$60) for doing the surveys listed above.

- You can get up to an additional \$225 for being a Peer Leader.
  - \$100 for participating in the training session

  - \$25 for recruiting your first friend to enroll in the study
     \$5 for each friend enrolled in the study after the first friend (Maximum of \$50) for up to 10 additional friends enrolled)
  - \$5 for each check-in online, in-person, or by text message (Maximum of \$50 for up to 10 check-ins).

Or

 You can earn up to 30 hours of community service for participating in the training, helping study staff to prepare for events (inventory, setup, and takedown), attending events, text message check ins, and recruiting other teens to enroll in the study.

If you choose academic volunteer service hours, you must follow the guidelines of your academic institutions to ensure the hours gained through AccessKCTeen 2.0 would count towards your overall requirement. If your academic institution does not allow volunteer hours from our study, you have the option to join the research study and earn up to \$225 (as listed above) for your participation

Problems or Questions? Please contact Melissa Miller (816) 302-1342 if you have any questions about this study. You may also call the Children's Mercy Hospitals' Pediatric Institutional Review Board (IRB) at (816) 731-7474 with questions or complaints about this study. The IRB is a committee that ensures that a research study is ethical and that the rights of study participants are protected.

Continuing with the study today means that you agree to be in AccessKCTeen 2.0 project.

